CLINICAL TRIAL: NCT04900116
Title: Comparison of Local Anesthetic Dose in PENG (Pericapsular Nerve Group) Block Performed for Postoperative Analgesia in Total Hip Replacement Operations
Brief Title: Comparison of Local Anesthetic Dose in PENG Block Performed in Total Hip Replacement Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nur Canbolat, Principal Investigator, M.D., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2020/1534
Record Dates: First submitted 2021-04-26; First posted 2021-05-25 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Pain, Postoperative
Keywords: Pericapsuler Nerve Group Block; Regional Anesthesia; Analgesic consumption; Postoperative analgesia; Numeric rating scale
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Injections; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): In this group, US guided PENG block will be performed with 20 ml 0.5% bupivacaine using a 22 gauge 10 mm block needle.
  Interventions: Drug: Bupivacaine HCl 0.5 % in 20 ML Injection
- Group 2 (Active Comparator): In this group, US guided PENG block will be performed with 20 ml 0.25% bupivacaine using a 22 gauge 10 mm block needle.
  Interventions: Drug: Bupivacaine HCl 0.25 % in 20 ML Injection
- Group 3 (Active Comparator): In this group, US guided PENG block will be performed with 20 ml 0.125% bupivacaine using a 22 gauge 10 mm block needle.
  Interventions: Drug: Bupivacaine HCl 0.125 % in 20 ML Injection
- Group 4 (Placebo Comparator): In this group, US guided PENG block will be performed with 20 ml saline solution (%0.9 NaCl) using a 22 gauge 10 mm block needle.
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Bupivacaine HCl 0.5 % in 20 ML Injection — In this group, US guided PENG block will be performed with 20 ml 0.5% bupivacaine using a 22 gauge 10 mm block needle.
  Other Names: Marcaine
  Arms: Group 1
Drug: Bupivacaine HCl 0.25 % in 20 ML Injection — In this group, US guided PENG block will be performed with 20 ml 0.25% bupivacaine using a 22 gauge 10 mm block needle.
  Other Names: Marcaine
  Arms: Group 2
Drug: Bupivacaine HCl 0.125 % in 20 ML Injection — In this group, US guided PENG block will be performed with 20 ml 0.125% bupivacaine using a 22 gauge 10 mm block needle.
  Other Names: Marcaine
  Arms: Group 3
Drug: NaCl 0.9% — In this group, US guided PENG block will be performed with 20 ml %0.9 NaCl solution using a 22 gauge 10 mm block needle (Control Group).
  Other Names: Saline Solution
  Arms: Group 4

SUMMARY:
The investigators research was designed as a single-center, prospective, randomized double-blind study. The patients undergoing total hip replacement surgery in Istanbul University Istanbul Medicine Faculty Department of Orthopedics and Traumatology will be included. Patients or persons who are legally authorized to make decisions on their behalf will be informed about the research and their written consent will be obtained. Patients who do not give consent will not be included in the study.

Patients will be given US guided PENG blocks using a 22 gauge 10 mm block needle after compliance with the rules of asepsia and antisepsis in the supine position according to the group of patients in which they were included.

PENG block will be done for postoperative analgesia. After the PENG block, a single dose of spinal anesthesia will be applied as a regional anesthesia method, in a sitting position, using the appropriate spinal needle, as is routinely applied in the investigators clinic. After the block is completed, the pinprick test will be done and the operation will be started after the successful completion of the block is confirmed. Oxygen will be given to the patients with a face mask at 4 lt / min throughout the operation. ECG, saturation, invasive / noninvasive blood pressure monitoring of the patients will be done. Measurements made at 5-minute intervals will be recorded.

In the investigators clinic, the use of PENG block and PCA (patient controlled analgesia) device with intravenous morphine for postoperative analgesia is routinely performed. In this study, four randomized groups will be formed together with the control group.

The local anesthetic solution given by the supervisor, whose doses of local anesthetic are predetermined (the investigators and participants do not know the dosage), with a total volume of 20 cc will be used. Local anesthetic agent will not be applied to the control group. As mentioned above, spinal anesthesia will be performed after PENG block and the operation will be started.

Pain score and total morphine consumption will be determined by visual pain scoring (VAS) at the postoperative 0, 6, 12, 24 and 48th hours by providing the use of a PCA device with intravenous morphine applied in routine practice to all four groups. As in routine practice, when VAS>4 after each interrogation, morphine 0.05 mg/kg iv will be administered as additional analgesia and the maximum will be increased to 10 mg. Pain management will continue when VAS <4.

DETAILED DESCRIPTION:
The investigators research was designed as a single-center, prospective, randomized double-blind study. After the approval of the Ethics Committee, the study will start and is aimed to be completed in 12 months.

The patients undergoing total hip replacement surgery in Istanbul University Istanbul Medicine Faculty Department of Orthopedics and Traumatology will be included. Patients or persons who are legally authorized to make decisions on their behalf will be informed about the research and their written consent will be obtained. Patients who do not give consent will not be included in the study.

Patients will be evaluated preoperative before surgery, a detailed history will be taken and physical examination will be carried out. Medical and surgical resume information will be obtained. Patients' Vas scores will be recorded before the operation. Patients will be taken to the operating room after premedication.

ECG, pulse oximeter, blood pressure monitoring will be performed in the operating room. Patients will be given US guided PENG blocks using a 22 gauge 10 mm block needle after compliance with the rules of asepsia and antisepsis in the supine position according to the group of patients in which they were included.

PENG block will be done for postoperative analgesia. After the PENG block, a single dose of spinal anesthesia will be applied as a regional anesthesia method, in a sitting position, using the appropriate spinal needle, as is routinely applied in the investigators clinic. After the block is completed, the pinprick test will be done and the operation will be started after the successful completion of the block is confirmed. Oxygen will be given to the patients with a face mask at 4 lt / min throughout the operation.

ECG, saturation, invasive / noninvasive blood pressure monitoring of the patients will be done. Measurements made at 5-minute intervals will be recorded.

In the investigators clinic, the use of PENG block and PCA (patient controlled analgesia) device with intravenous morphine for postoperative analgesia is routinely performed. In this study, four randomized groups will be formed together with the control group. Computer-generated random numbers will be used for simple randomization of patients.

The local anesthetic solution given by the supervisor, whose doses of local anesthetic are predetermined (the investigators and participants do not know the dosage), with a total volume of 20 cc will be used. Local anesthetic agent will not be applied to the control group. As mentioned above, spinal anesthesia will be performed after PENG block and the operation will be started.

Pain score and total morphine consumption will be determined by visual pain scoring (VAS) at the postoperative 0, 6, 12, 24 and 48th hours by providing the use of a PCA device with intravenous morphine applied in routine practice to all four groups. As in routine practice, when VAS>4 after each interrogation, morphine 0.05 mg/kg iv will be administered as additional analgesia and the maximum will be increased to 10 mg. Pain management will continue when VAS <4.

Patients are followed up in the service for 48 hours postoperatively in routine practice. In the postoperative period, patients will be evaluated in terms of additional nausea and vomiting, first mobilization time, hospitalization time, amount of morphine consumed and additional analgesic need, onset time of narcotic analgesic need, preoperative and postoperative in the first month Depression-BECK Score, quadriceps weakness, postop patient satisfaction and surgical satisfaction. During the procedure, complications such as failed block, nerve damage, vascular injury, intravenous injection of local anesthetic, local anesthetic toxicity and allergic reactions will be recorded.

Before the study, it was determined that at least 84 patients should be collected in the power analysis performed with the help of similar literature data. After collecting the demographic data and morphine consumption data of the patients, the data will be transferred to the statistical program called SPSS and statistical analysis will be made.The investigators study does not contain any modifications other than the investigators daily routine practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total hip replacement surgery under regional anesthesia
* ASA(American Society of Anesthesiology) 1-3
* Receiving consent that accept regional analgesia

Exclusion Criteria:

* Refusal of regional anesthesia
* Infection on the local anesthetic application area
* Infection in the central nervous system
* Coagulopathy
* Increased intracranial pressure (Brain tumors)
* Known allergy against local anesthetics
* Anatomical difficulties

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (0-10) pain scores for patients | Up to 48 hours
  The VAS (Visual Analog Scale, 0 mm ''no pain'', to 100 mm, ''the worst pain possible'')

SECONDARY OUTCOMES:
Opioid (mg) consumption | during surgery and postoperative period up to 48th hours.
  Opioid (mg) consumption
Time of onset of narcotic analgesic need | during surgery and postoperative period up to 48th hours.
  (If VAS > 4, morphine 0.05 mg/kg IV will be administered as rescue analgesia additional analgesia and maximum will be increased to 10 mg.
Incidence of side effects | during surgery and postoperative period up to 48th hours.
  Incidence of nausea and vomiting
Incidence of quadriceps weakness | postoperative period up to 48th hours and postoperative in the first month
  Physical examination for lower extremity
Time until postoperative first mobilization | Up to 48 hours
  First mobilization time
Length of hospital stay | Through study completion, an average of 1 week
  Hospitalization
Beck depression inventory scores | Will be done 3 times 1- on pre-operative hospitalization 2- in the hospital after surgery 3- in the 1st month follow-up after surgery
  (1-10 These ups and downs are considered normal, 11-16 Mild mood disturbance, 17-20 Borderline clinical depression, 21-30 Moderate depression, 31-40 Severe depression, Over 40 Extreme depression)
Patient satisfaction | postoperative period up to 48th hours and postoperative in the first month
  Satisfaction score; 0- very unsatisfied, 3- very satisfied
Surgeon satisfaction | postoperative period up to 48th hours and postoperative in the first month
  Satisfaction score; 0- very unsatisfied, 3- very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: İlke Akay Akgül, MD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Result] Abdalrahim MS, Majali SA, Stomberg MW, Bergbom I. The effect of postoperative pain management program on improving nurses' knowledge and attitudes toward pain. Nurse Educ Pract. 2011 Jul;11(4):250-5. doi: 10.1016/j.nepr.2010.11.016. Epub 2010 Dec 24. PMID 21186139
- [Result] Krishna Prasad GV, Khanna S, Jaishree SV. Review of adjuvants to local anesthetics in peripheral nerve blocks: Current and future trends. Saudi J Anaesth. 2020 Jan-Mar;14(1):77-84. doi: 10.4103/sja.SJA_423_19. Epub 2020 Jan 6. PMID 31998024
- [Result] Bilal B, Oksuz G, Boran OF, Topak D, Dogar F. High volume pericapsular nerve group (PENG) block for acetabular fracture surgery: A new horizon for novel block. J Clin Anesth. 2020 Jun;62:109702. doi: 10.1016/j.jclinane.2020.109702. Epub 2020 Jan 9. No abstract available. PMID 31927234
- [Result] Aksu C, Cesur S, Kus A. Pericapsular Nerve Group (PENG) block: Controversial points about anatomical differences. J Clin Anesth. 2020 May;61:109701. doi: 10.1016/j.jclinane.2020.109701. Epub 2020 Jan 8. No abstract available. PMID 31924520